CLINICAL TRIAL: NCT04984811
Title: A Multicenter, Open-label, Single-arm Phase II Study to Evaluate Anti-tumor Efficacy and Safety of NT-I7 in Combination With Atezolizumab in Subjects With Previously Untreated, PD-L1-expressing, Locally Advanced or Metastatic NSCLC
Brief Title: NT-I7 in Combination With Atezolizumab in Previously Untreated, PD-L1-expressing, Locally Advanced or Metastatic NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NeoImmuneTech (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIT-119
Record Dates: First submitted 2021-07-14; First posted 2021-08-02 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Non-Small Cell Lung Cancer; Non-Small Cell Lung Carcinoma; Nonsmall Cell Lung Cancer; Non Small Cell Lung Cancer
Keywords: Advanced; Metastatic; NSCLC; PD-L1; Atezolizumab; NT-I7; Non Small Cell Lung Cancer; Non-small Cell Lung Cancer; Non-Small Cell Lung Carcinoma; Nonsmall Cell Lung Cancer; efineptakin alfa; efineptakin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — efineptakin alfa; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NT-I7 and atezolizumab (Experimental): Participants with no prior systemic therapy for advanced NSCLC will receive 1200 μg/kg NT-I7 IM on Day 1 and every 6 weeks and atezolizumab IV 1200 mg every 3 weeks until disease progression.
  Interventions: Drug: efineptakin alfa; Drug: Atezolizumab

INTERVENTIONS:
Drug: efineptakin alfa — 1200 μg/kg NT-I7 administered intramuscularly (IM) once every 6 weeks (Q6W) starting on Cycle 1. The treatment will be continued up to a maximum of 35 cycles (approximately 2 years).
  Other Names: NT-I7
Drug: Atezolizumab — 1200 mg atezolizumab administered intravenously (IV) once every 3 weeks (Q3W) starting on Cycle 1. The treatment will be continued up to a maximum of 35 cycles (approximately 2 years).
  Other Names: Tecentriq

SUMMARY:
This is a multicenter, open-label, single-arm Phase II study to evaluate anti-tumor efficacy and safety of NT-I7 in combination with atezolizumab in subjects with PD-L1-expressing (TPS ≥ 1%), metastatic (Stage IV) or locally advanced squamous or non-squamous NSCLC who have not received prior systemic therapy in the metastatic or locally advanced setting. Eligible subjects must have measurable disease according to RECIST 1.1. This Phase II study will enroll up to 83 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed metastatic or locally advanced NSCLC, and have not received prior systemic therapy. Subjects with locally advanced disease must have Stage III NSCLC and are not candidates for surgical resection or definitive chemoradiation
* Tumor PD-L1 expression (TPS≥1%) as determined by PD-L1 22C3 immunohistochemistry local or central assay.
* Have measurable disease
* Agree to provide screening biopsy (or archival tissue) at screening to assess PD-L1
* ECOG 0-1
* Adequate hematologic and end organ function

Exclusion Criteria:

* Prior systemic anti-cancer therapy
* NSCLC with EGFR, or ALK, or BRAF or ROS or RED or other genomic tumor aberrations which have available therapy
* Prior radiotherapy within 2 weeks of start of study treatment
* Known active CNS metastasis or carcinomatous meningitis
* Severe reactions to mAbs or IV immunoglobulin preparations
* Autoimmune disease history in past two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | approximately 2 years
  The percentage of subjects with a best overall response (BOR) of a complete response (CR) or partial response (PR), per RECIST 1.1 and iRECIST as determined by the investigator.

SECONDARY OUTCOMES:
Duration of response (DoR) | approximately 2 years
  Time from the first occurrence of a documented objective response to the time of the first documented disease progression or death from any cause, whichever occurs first, per RECIST 1.1 and iRECIST as determined by the investigator.
Disease Control Rate (DCR) | approximately 2 years
  The proportion of subjects with a best overall response of CR, PR or SD, per RECIST 1.1 and iRECIST as determined by the investigator.
Progression Free Survival (PFS) | approximately 2 years
  The time from the first study treatment (Cycle 1, Day 1) to the first occurrence of progression or death from any cause, whichever occurs first, per RECIST 1.1 and iRECIST as determined by the investigator.
Overall survival (OS) | approximately 2 years
  The time from first study treatment (Cycle 1, Day 1) to death from any cause.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - University of South Alabama, Mobile, Alabama
  - TOI Clinical Research, Cerritos, California
  - Eastern CT Hematology & Oncology Associates, Norwich, Connecticut
  - Florida Cancer Specialists - South Research Office, Fort Myers, Florida
  - BRCR Medical Center, Plantation, Florida
  - Florida Cancer Specialists - North Research Office, St. Petersburg, Florida
  - Florida Cancer Specialists - East Research Office, West Palm Beach, Florida
  - University Cancer and Blood Center, Athens, Georgia
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Pikeville Medical Center, Inc., Pikeville, Kentucky
  - MaineHealth Cancer Care, South Portland, Maine
  - TidalHealth Peninsula Regional, Inc., Salisbury, Maryland
  - Summit Health Medical Center, Florham Park, New Jersey
  - East Carolina University, Greenville, North Carolina
  - Zangmeister Cancer Center, Columbus, Ohio
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Tennessee Oncology - Chattanooga, Chattanooga, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Tennessee Oncology - Nashville, Nashville, Tennessee
  - Renovatio Clinical - El Paso, El Paso, Texas
  - Renovatio Clinical - The Woodlands, The Woodlands, Texas